CLINICAL TRIAL: NCT04848311
Title: Indocanine Green as Tracer for Lymph Nodes Dissection in Station 253 of Rectal and Sigmoid Colon Carcinoma
Brief Title: Indocanine Green as Tracer for Lymph Nodes Dissection in Station 253
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NFEC-2021-073
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2020-12

CONDITIONS: Rectal Carcinoma; Sigmoid Colon Carcinoma
Keywords: ICG; 253 lymph nodes; rectal carcinoma; sigmoid colon carcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG group (Experimental): Patients in the ICG group will undergo endoscopic injection of ICG 4 hours before surgery. The ICG powder will be dissolved in 2.5mg/ml of sterile water. ICG will be injected along the submucosa at 4 points around the primary tumor,for a total volume of 10ml.
  Interventions: Procedure: lymph nodes dissection at 253 station assisted by ICG
- CLgroup (No Intervention): Patients in the CL group will undergo routine laparoscopic lymph nodes dissection instead of using any tracer.

INTERVENTIONS:
Procedure: lymph nodes dissection at 253 station assisted by ICG — In ICG group :All patients will be subjected to laparoscopic radical resection with station 253 lymph nodes dissection by fluorescence laparoscopic.
  Arms: ICG group

SUMMARY:
This is a prospective randomized controlled study. investigators will randomly assign patients to the indocanine green (ICG) group and control (CL)group to compare the differences of lymph nodes dissection in station 253 between the two groups.

DETAILED DESCRIPTION:
ICG is a registered and FDA-approved non-specific fluorescent probe for optical imaging in clinical settings. The properties of ICG ,which is a water-soluble amphiphilic molecule with a molecular weight of 775 Dalton and a hydrodynamic diameter of 1.2nm ,render it an excellent lymphatic contrast agents if injected into the lymphatic system. ICG near-infrared(NIR) fluorescent imaging has achieved satisfactory results in the localization of sentinel lymph nodes in patients with breast cancer,non-small cell lung cancer,and gastric cancer. Liang et al have suggested that 253 lymph nodes dissection in rectal cancer is technically demanding ,and that learning curve for laparoscopic 253 lymph nodes dissection requires minimally 20 procedures. Currently,it was still controversial about 253 lymph nodes dissection in rectal cancer surgery. However, lymph node involvement is a major prognostic factor for survival after rectal cancer surgery. Therefore, it is necessary to harvest more station 253 nodes for the better long-term survival and the more precise staging.

In this study, investigators will randomly assign patients to the indocanine green (ICG) group and control (CL)group. Number of harvested station 253 lymph nodes, number of positive station 253 lymph nodes, will be evaluated and compared. Investigators will also evaluate patients, operative time, blood loss, post-operative hospital stay and complications.

ELIGIBILITY:
Inclusion Criteria:

(1)18-80 years of age (2)American Society of Anesthesiologists (ASA) class 1-3 (3)single rectal or sigmoid colon carcinoma confirmed pathologically by endoscopic biopsy (4)planned laparoscopic radical resection (5)Written informed consent

Exclusion Criteria:

1. previous abdominal tumor surgery
2. women who are pregnant or breast feeding
3. emergency patients with obstruction or perforation
4. T4b cancer evaluated by CT or MRI or endoscopic ultrasonography
5. pelvic or distant metastasis
6. T1 cancer planned local excision
7. allergic constitution patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
number of harvested station 253 lymph nodes | one week after operation
  number of harvested station 253 lymph nodes,number of positive station 253 lymph nodes,rate of positive station 253 lymph nodes

SECONDARY OUTCOMES:
number of harvested station 251 lymph nodes | one week after operation
  number of harvested station 251 lymph nodes, number of positive station 251 lymph nodes, rate of positive station 251 lymph nodes,
number of harvested station 252 lymph nodes | one week after operation
  number of harvested station 252 lymph nodes, number of positive station 252 lymph nodes , rate of positive station 252 lymph nodes
number of total lymph nodes harvested | one week after operation
  number of total lymph nodes harvested, number of total positive lymph nodes ,rate of total positive lymph nodes

OTHER OUTCOMES:
operative time | intraoperative
post-operative data | one hour after operation
  blood loss
post-operative hospital stay | two weeks after operation
  post-operative hospital stay
complications | two weeks after operation
  post-operative data

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yan, M.D,Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wan J, Wang S, Yan B, Tang Y, Zheng J, Ji H, Hu Y, Zhuang B, Deng H, Yan J. Indocyanine green for radical lymph node dissection in patients with sigmoid and rectal cancer: randomized clinical trial. BJS Open. 2022 Nov 2;6(6):zrac151. doi: 10.1093/bjsopen/zrac151. PMID 36515673